CLINICAL TRIAL: NCT03455101
Title: Turkish Nationwide SurvEy of Glycemic and Other Metabolic Parameters of Patients With Diabetes Mellitus (TEMD Study)
Brief Title: Turkish Nationwide SurvEy of Glycemic and Other Metabolic Parameters of Patients With Diabetes Mellitus
Acronym: TEMD
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Alper Sonmez, Prof. Dr., Gulhane School of Medicine
Other Study IDs: GSM012017
Record Dates: First submitted 2017-09-24; First posted 2018-03-06 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-02

CONDITIONS: Diabetes Mellitus
Keywords: Cardiovascular risk status; Optimal metabolic control
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with diabetes mellitus: Patients with type 1 or type 2 diabetes who were under follow-up in the same center for at least a year.
  Interventions: Other: There is no intervention.

INTERVENTIONS:
Other: There is no intervention. — There is no intervention.

SUMMARY:
This study evaluates the overall cardiovascular risk status and best predictors of optimal metabolic control of Turkish adult patients with diabetes mellitus.

DETAILED DESCRIPTION:
Diabetes mellitus is one of the most common chronic diseases with an increasing prevalence worldwide.The prevalence of diabetes is also increased significantly in Turkey, from 7.2 % in 2002 to 13.7% in 2012.This increasing prevalence leads to serious public health problems and a significant economic burden. Therefore, the optimal treatment of diabetes and prevention of diabetic complications, especially the cardiovascular outcomes, is utmost important. Although achieving glycemic targets in patients with diabetes is of great importance, blood glucose is not the only predictor of cardiovascular outcome in diabetes. Optimization of other metabolic parameters such as lipids, arterial blood pressure (ABP), and body weight as well as a healthy lifestyle are utmost important. As there is hardly enough data about glycemic and other metabolic control parameters in Turkish adult patients with type 1 or type 2 diabetes, this nationwide survey was performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 or type 2 diabetes
* Upper than 18 years old
* To be under follow-up in the same center for at least one year.

Exclusion Criteria:

* Pregnancy
* Younger than 18 years old,
* History of decompensated liver disease,
* History of psychiatric disorders interfering cognition or compliance
* History of bariatric surgery
* History of renal replacement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 or type 2 diabetes who were under follow-up in the same tertiary endocrine unit for at least a year were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 5240 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Glycemia control status of Turkish adult patients with diabetes mellitus | 7 days
  Glycemia control will be defined as good control if the mean HbA1c level of patients < 7% or poor control if the mean HbA1c level of patient > 7%

SECONDARY OUTCOMES:
Blood pressure control status of Turkish adult patients with diabetes mellitus | 7 days
  Home blood pressure <135/85 mmHg will be defined as under control.
Lipid control status of Turkish adult patients with diabetes mellitus. | 7 days.
  Triglyceride < 150 mg/dl, LDL-C < 100 mg/dl, HDL-C > 40 mg/dl for men, and HDL-C > 50 mg/dl for women will be defined as under control.
Weight control status of Turkish adult patients with diabetes mellitus. | 7 days.
  Body mass index < 30 kg/m2 will be defined as under control. Weight and height will be combined to report body mass index in kg/m2.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane School of Medicine Department of Endocrinology and Metabolism, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sonmez A, Tasci I, Demirci I, Haymana C, Barcin C, Aydin H, Cetinkalp S, Ozturk FY, Gul K, Sabuncu T, Satman I, Bayram F; TEMD Study Group. A Cross-Sectional Study of Overtreatment and Deintensification of Antidiabetic and Antihypertensive Medications in Diabetes Mellitus: The TEMD Overtreatment Study. Diabetes Ther. 2020 May;11(5):1045-1059. doi: 10.1007/s13300-020-00779-0. Epub 2020 Feb 22. PMID 32088879